CLINICAL TRIAL: NCT03050255
Title: Short-term Effects of Supplemental Oxygen During Walking in Hypoxemic Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Short-term Effects of Supplemental Oxygen in Patients With IPF
Acronym: IPFO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Linde AG (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr., Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IPF-O2-Study
Record Dates: First submitted 2016-11-25; First posted 2017-02-10 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: supplemental oxygen; walking capacity; exercise capacity; endurance shuttle walk test
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Air; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ESWT order 1 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. medical air (MA)
  2. Oxygen (2 Liter/min)
  3. Oxygen (4 Liter/min)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)
- ESWT order 2 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. medical air (MA)
  2. Oxygen (4 Liter/min)
  3. Oxygen (2 Liter/min)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)
- ESWT order 3 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. Oxygen (2 Liter/min)
  2. Medical air (MA)
  3. Oxygen (4 Liter/min)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)
- ESWT order 4 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. Oxygen (2 Liter/min)
  2. Oxygen (4 Liter/min)
  3. Medical air (MA)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)
- ESWT order 5 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. Oxygen (4 Liter/min)
  2. Medical air (MA)
  3. Oxygen (2 Liter/min)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)
- ESWT order 6 (Experimental): Subject performs endurance shuttle walk tests (ESWT) under following conditions in the following order:
  1. Oxygen (4 Liter/min)
  2. Oxygen (2 Liter/min)
  3. Medical air (MA)
  Interventions: Other: Medical air; Other: Oxygen (2Liter/min); Other: Oxygen (4Liter/min)

INTERVENTIONS:
Other: Medical air
Other: Oxygen (2Liter/min)
Other: Oxygen (4Liter/min)

SUMMARY:
Although exercise-induced desaturation is frequently observed in patients with idiopathic pulmonary fibrosis (IPF) short-term effects of supplemental oxygen during walking have not been investigated yet. Given, that walking ability is the most important activity of daily life, the aim of our study is to investigate the effects of supplemental oxygen on endurance walking capacity in hypoxemic IPF patients. In this study patients will perform 3 endurance shuttle walk tests (ESWTs) at 85% of their individual peak performance using medical air (=compressed room air, 2 liters/minute), 2 liters/minute oxygen, 4 liters/minute Oxygen in a double-blinded fashion and random order.

Since there are only limited pharmacological treatment options for IPF patients, this study may help to provide novel information about the short-term effects of supplemental oxygen. Furthermore it may help to investigate possibilities to optimize oxygen therapy in order to facilitate patients´ participation in activities of daily life and not at least to improve patients´ quality of life.

DETAILED DESCRIPTION:
Rationale:

Exercise-induced desaturation is frequently observed in patients with idiopathic pulmonary fibrosis and predicts poorer outcomes. However, prospective studies with larger sample sizes and those investigating the effect of oxygen on endurance time, oxygen saturation and breathing frequency during walking are lacking. Given that walking is the most important activity of daily life to preserve the maintenance and to participate in social life, we aim to investigate the effects of supplemental oxygen during walking in IPF patients.

The endurance shuttle walk test (ESWT) is a well validated test with high reliability and validity for measuring endurance walking capacity in patients with chronic obstructive pulmonary disease (COPD). The advantage of this test in contrast to the 6-minute walk test is that the ESWT is performed at 85% of the individual maximum that is close to the intensity of typical daily activities. Additionally, by using the ESWT it is possible to determine the maximum duration of exercise and to compare values at isotime (= time point when the shortest of the 3 ESWTs ends), whereas values at the end of different six-minute walk tests (6MWTs) are not comparable in case of different distances.

Aim:

To investigate the short-term effects of supplemental oxygen on endurance capacity during walking (ESWT) in patients with idiopathic pulmonary fibrosis.

Design:

This study is a randomized, controlled, double-blinded cross-over trial. Following an initial incremental shuttle walk test (ISWT) in order to determine the individual maximum walking capacity, patients will perform 3 endurance shuttle walk tests (ESWT) at 85% of the maximal pace. In randomized order, patients will complete one ESWT on 2l/min oxygen, one on 4l/min oxygen and one on medical air (=compressed room air), whereas the patients as well as the investigator will be blinded to the gas mixture provided. All 3 conditions will be provided via nasal cannula. The time between the two ESWTs will be 24 hours in order to give enough time for regeneration. Endurance Walking capacity as measured by the ESWT will be used as the primary outcome.

ELIGIBILITY:
Inclusion criteria:

* patients with idiopathic pulmonary fibrosis and hypoxemia at rest or during exercise (PaO2 <55 mmHg or SpO2 <88%)
* Written informed consent

Exclusion criteria:

* Forced vital capacity < 50% pred.
* Clinical signs of any cardial comorbidity
* Not able to walk
* Oxygen flow needed during exercise > 4l/min

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Endurance time (in seconds) measured by endurance shuttle walk test | Time until Patient terminates ESWT due to leg fatigue or dyspnea, up to 20 minutes

SECONDARY OUTCOMES:
Change of breathing frequency during endurance shuttle walk test | change from baseline to the end of the ESWT, up to 20 minutes
  measured by NOX-T3 (NoxMedical, Reykjavik, Iceland)
Change of Oxygen saturation during endurance shuttle walk test | change from baseline to the end of the ESWT, up to 20 minutes
  continuous transcutaneous recording during endurance shuttle walk test via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of heart rate during endurance shuttle walk test | change from baseline to the end of the ESWT, up to 20 minutes
  continuous transcutaneous recording during endurance shuttle walk test via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of partial pressure of carbon dioxide during endurance shuttle walk test | Change from baseline to the end of the ESWT, up to 20 minutes
  continuous transcutaneous recording during endurance shuttle walk test via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of inspiratory capacity during endurance shuttle walk test | Change from baseline to the end of the ESWT, up to 20 minutes
  measured by Spiropalm 6MWT (Cosmed, Italy)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof., Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Undecided